CLINICAL TRIAL: NCT06221956
Title: Effectiveness of a Digital Health Application for Subacute and Chronic Back Pain (Relevis): a Randomized Controlled Trial
Brief Title: Effectiveness of a Digital Health Application for Subacute and Chronic Back Pain (Relevis)
Acronym: APRICOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gaia AG (Industry)
Collaborators: University Hospital Schleswig-Holstein (Other); Philipps Universität Marburg (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: relevis RCT 2024
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- relevis + TAU (Experimental): Participants allocated to the intervention group will receive access to relevis in addition to treatment as usual (TAU).
  relevis is a digital health application designed for individuals with subacute or chronic back pain, accessible through a web browser. The application consists of six physical exercise modules that cover four exercises with thiree different levels of difficulty, each, and ten interactive "conversations" on different topics (changes in the body, pain development and processing, chronic pain, pain and mood, relaxation and mindfulness, becoming active against pain, stress and pain, nutrition and pain, sleep and pain, work and pain). "Conversations" are accompanied by illsutrations, audio recordings, motivating text messages, worksheets, and summaries. Users are also encouraged to regularly complete short questionnaires to monitor their complaints. Once registered, the program remains accessible for 180 days.
  Interventions: Behavioral: relevis
- TAU (No Intervention): Participants allocated to the control group will receive access to treatment as usual (TAU).

INTERVENTIONS:
Behavioral: relevis — Participants will receive access to the digital health intervention relevis in addition to TAU.
  Arms: relevis + TAU

SUMMARY:
This clinical trial with 276 patients with subacute or chronic back pain aims to investigate the effectiveness of the unguided digital therapeutic relevis for patients with subacute or chronic back pain. Inclusion criteria are: age ≥ 18 years, presence of subacute (6-12 weeks) or chronic (>12 weeks) back pain, attested by a medical certificate (relevant ICD-10-GM diagnoses: M47.8x, M47.9x, M54.5, M54.8x, M54.9x, M51.0x, M51.1x, M51.2), impaired functional ability [Oswestry Disability Index (ODI) ≥ 21], consent to participation, sufficient knowledge of the German language. Exclusion criteria are: change in treatment of back pain in the past month, planned change in treatment of back pain in the next 3 months, prior use of other online programs/apps for back pain, history of back, hip or knee surgery in the past 6 months, history of more than one back surgery in lifetime, presence of a specific cause for back pain (e.g., fracture, infection, neuropathies [except when due to disc prolapse], axial spondyloarthritis), tumor or metastases, cauda equina syndrome, acute myocardial infarction, unstable coronary heart disease/angina pectoris or heart failure, acute thrombosis, manifest osteoporosis, acute fevers, rheumatic autoimmune diseases.

Patients will be randomized and allocated to either an intervention group in a 1:1 ratio, in which they will receive access to relevis in addition to treatment as usual (TAU, n = 138), or to a control group, in which they will receive only TAU (n = 138). TAU is defined as any therapy prescribed or recommended by the GP or specialists (e. g. orthopedic surgeon, rheumatologists etc.) which may include physiotherapy, injections in the spine, drug therapy, orthesis, etc. (1,2). The primary endpoint will be the functional impairment, measured by the ODI, with three months post-allocation being the primary time point for assessment of effectiveness (T1). Six months post-allocation (T2) will be used as the follow-up assessment endpoint. Secondary endpoints will be depression, work and social functioning, pain intensity, and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Presence of subacute (6-12 weeks) or chronic (>12 weeks) back pain
* Submission of a medical certificate attesting to the presence of at least one of the following ICD-10-GM diagnoses of back pain:

  * M47.8x - Spondylosis
  * M47.9x - Other spondylosis
  * M54.5 - Back pain
  * M54.8x - Other back pain
  * M54.9x - Unspecified back pain
  * M51.0x - Thoracic, thoracolumbar and lumbosacral intervertebral disc disorders with myelopathy
  * M51.1x - Thoracic, thoracolumbar and lumbosacral intervertebral disc disorders with radiculopathy
  * M51.2 - Other thoracic, thoracolumbar and lumbosacral intervertebral disc displacement
* Impaired functional ability (ODI ≥ 21)
* Consent to participate
* Sufficient knowledge of the German language

Exclusion Criteria:

* Change in treatment of back pain in the past month
* Planned change in treatment of back pain in the next 3 months
* Prior use of other online programs/apps for back pain
* History of back, knee or hip surgery in the past 6 months
* History of more than one back surgery during lifetime
* Presence of a specific cause for back pain, e.g.:

  * Fracture
  * Infection
  * Neuropathies (except when due to disc prolapse)
  * Axial spondyloarthritis
* Tumor or metastases
* Cauda equina syndrome
* Acute myocardial infarction
* Unstable coronary heart disease/angina pectoris or heart failure
* Acute thrombosis
* Manifest osteoporosis
* Acute fevers
* Rheumatic autoimmune diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2025-01-23 (Estimated); Study Completion 2025-01-23 (Estimated)

PRIMARY OUTCOMES:
Functional Impairment | 3 months
  Oswestry Low Back Pain Disability Questionnaire (ODI). Total score ranging from 0-100; higher scores mean higher functional impairment (worse outcome).

SECONDARY OUTCOMES:
Depressive Symptomatology | 3 months
  Patient Health Questionnaire (PHQ-9). Total score ranging from 0-27; higher scores mean higher depressive symptomatology (worse outcome).
Work and Social Functioning | 3 months
  Work and Social Adjustment Scale (WSAS). Total score ranging from 0-40; higher scores mean higher disability (worse outcome).
Intensity of Back Pain | 3 months
  Numeric Rating Scale (NRS). Score ranging from 0-10; higher scores mean higher pain (worse outcome).
Health-related Quality of Life | 3 months
  Assessment of Quality of Life - 8 Dimensions (AQoL-8D). Total score ranging from 0-100; higher scores mean higher quality of life (better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Kamila Jauch-Chara, MD, Principal Investigator — University Hospital Schleswig-Holstein
Locations (1):
- GAIA AG, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No